CLINICAL TRIAL: NCT00716365
Title: USF Hemostasis: USage of HemCon for Femoral Hemostasis After Percutaneous
Brief Title: USF Hemostasis: USage of HemCon for Femoral Hemostasis After Percutaneous Procedures
Acronym: USF-Hemostasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Meir Medical Center (Other)
Responsible Party: Prof. Morris Mosseri, Division of Cardiology, Meir Medical Center, Kfar-Saba, Israel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0152-07MMC
Record Dates: First submitted 2008-05-22; First posted 2008-07-16 (Estimated); Last update posted 2011-08-16 (Estimated); Status verified 2011-08

CONDITIONS: Coronary Angiography
Keywords: angiography; hemostasis; femoral artery; duplex

ARMS (1):
- HemCon (Experimental): The purpose of this trial is to test HemCon pad after diagnostic percutaneous coronary angiography as an adjunct to manual compression to better control vascular access site bleeding and reduce time-to-hemostasis.
  The HemCon bandage (containing a carbohydrate called chitosan, found in the shells of shrimp, lobster and beetles) will be used to shorten the time needed to achieve hemostasis, time to patient's ambulation, and patient's.
  Interventions: Device: HemCon bandage

INTERVENTIONS:
Device: HemCon bandage — 5 cm X 5 cm
  Other Names: HemCon

SUMMARY:
USF Hemostasis - USage of HemCon for Femoral Hemostasis after Percutaneous Procedures. A Comparative Open Label Study The purpose of this trial is to test HemCon pad after diagnostic percutaneous coronary angiography as an adjunct to manual compression to better control vascular access site bleeding and reduce time-to-hemostasis.

We hypothesize that the use of HemCon bandage (containing a carbohydrate called chitosan, found in the shells of shrimp, lobster and beetles) will shorten the time needed to achieve hemostasis, time to patient's ambulation, and patient's satisfaction without increasing vascular complications.

278 patients undergoing diagnostic coronary angiography receiving 2500 u intravenous Heparin will be studied and randomized for manual homeostasis with either a HemCon or a regular pad. Primary efficacy endpoint will be time to hemostasis. Secondary endpoints will be safety (complication rate) and satisfaction of patients regarding time to sitting incline and time to ambulation. 25% of patients from each arm will be randomized for Duplex examination of the femoral artery at the access site.

DETAILED DESCRIPTION:
USF Hemostasis USage of HemCon for Femoral Hemostasis after Percutaneous Procedures A Comparative Open Label Study Introduction After completion of angiography performed via the femoral artery, hemostasis is achieved by applying local pressure either manually or by mechanical devices for 10-20 minutes. This is time consuming for the physician, uncomfortable for the patient and occasionally complicated with vascular events that increase morbidity and hospital duration and reduce patient satisfaction. Closure devices have been developed to shorten pressure time but they are costly.

The HemCon pad is composed of a bandage containing a carbohydrate called chitosan, found in the shells of shrimp, lobster and beetles. Its molecules are positively charged and attract the negatively charged blood cells and platelets, and thus promote clotting. Chitosan hemorrhage control dressings have been shown to be effective in animal models of severe hemorrhage (1-4). Bandage. U.S. military personnel in the Iraquean and Afghanistan conflicts have used the HemCon Bandage to successfully stop arterial hemorrhage not controlled by conventional bandages in more then 64 patients without adverse effects (3,5). The HemCon bandage is also an FDA-cleared hemostatic dressing suitable for use in hemodialysis access puncture (2).

The purpose of this trial is to test HemCon pad after diagnostic percutaneous coronary angiography as an adjunct to manual compression to better control vascular access site bleeding and reduce time-to-hemostasis.

We hypothesize that the use of HemCon bandage will shorten the time needed to achieve hemostasis, time to patient's ambulation, and patient's satisfaction without increasing vascular complications.

Endpoints Primary endpoint

* Compare efficacy (time to hemostasis) of HemCon to regular pads Secondary endpoints
* Compare efficacy (time to ambulation) of HemCon to regular pads
* Compare safety (complication rate) of HemCon to regular pads using a protocol of shorter time to ambulation with the HemCon pad.
* Compare satisfaction of patients regarding time to sitting incline and time to ambulation.

Patients 278 patients undergoing diagnostic coronary angiography receiving 2500 u intravenous Heparin will be studied and randomized as written hereinafter.

Inclusion Criteria:

* Age 18-80 years old
* Signing an informed consent
* Percutaneous coronary angiography with a 6 french sheath via the femoral artery
* Post catheterization non-invasive systolic blood pressure 150 mm Hg

Exclusion criteria:

* STEMI
* Patients who received IIb-IIIa antagonists before or during angiography.
* Patients who received more than 2500u IV Heparin or more than 0.5 mg/kg LMWH within 8 hours before the procedure.
* Known bleeding tendency, disturbed clotting system or platelet function
* Evidence of bleeding or hematoma at the access site prior to sheath removal.

Protocol

Heparin treatment:

All patients will receive IV 2500 u Heparin immediately after introducing the femoral sheath.

* Procedure duration:

Procedure duration will be recorded in minutes.

* Randomization:

A 1:1 randomization of HemCon and regular pad will be performed after completion of the procedure. Envelopes marked with consecutive numbers will contain a note written: "HemCon pad" or "Regular pad ". Notes content will be randomized by a computer program.

After the procedure is completed and a decision is taken to withdraw the sheath the next consecutive envelope will be opened to determine the sheath removal technique to be used.

* Arterial sheath removal:

  1. The femoral sheath will be removed at the patient's bed (and not on the angiography table). One ml of blood will be allowed to flow from the access site. A HemCon or a regular pad (according to randomization) will be applied manually with occlusive pressure for 5 minutes.
  2. After 5 minutes the operator will release the pressure. If bleeding continues, application of local pressure will be resumed. After this stage, the operator is allowed to release the pressure after every 5 minutes or longer at the operator's discretion. The total numbers of pressure release and the total time to hemostasis will be recorded.
  3. After achieving hemostasis a pressure bandage will be applied at the access site for 3 hours.

     Bed rest:

  <!-- -->

  1. Minimal bed rest duration will be 2 hours. Longer bed rest duration in increments of 30 minutes will be decided at the operator's discretion according to hemostasis. Total bed rest time will be recorded.
  2. During bed rest the operator may allow the patient to sit up in 450 incline after 1 hour. Time to sitting up will be recorded.
  3. If hematoma occurs, it will be evaluated by palpation and diameter measurement will be recorded.
* Ambulation:

After bed rest, ambulation is allowed providing no confounding events such as blood pressure abnormalities and hematoma have developed.

* In hospital follow-up:

  1. A duplex examination of the femoral artery at the access site will be performed at the operator's discretion.
  2. One day after the procedure patient's complaints and physical findings will be recorded.
  3. Blood count will be taken from all patients on the day after the procedure. Earlier blood count and other blood examinations may be taken at the operator's discretion and will be recorded.
* Discharge:

The patient will be discharged at the operator's discretion. Complications or adverse events will be noted and recorded upon discharge.

• Out of hospital and patient's satisfaction follow up: One day after discharge the patient will be contacted by phone and asked for any procedural complications (groin pain, hematoma) that appeared after discharge. If needed, the patient will be invited to the hospital for further investigation.

During the phone call the patient will be asked of his / her satisfaction of the ambulation procedure at a scale of 1-10 (10 mostly satisfactory).

Statistics

The following data will be compared between the 2 groups using t-test:

* Time to hemostasis
* Duration of bed rest (total, supine position and incline sit-up position)
* Incidence of minor and major hematoma
* Hematoma size
* Post procedural stay at the hospital
* Level of satisfaction evidenced in post-procedure satisfaction surveys. The number of patients to be studied (278) was calculated with the assumption that the HemCon will achieve a decrease of 30% in hemostasis time (the primary endpoint), with alpha value of 0.05 and power of 0.8.

REFERENCES

1. Pausateri AE, McCarthy SG, et al. Effect of chitosan-based hemostatic dressing on blood loss and survival in a model of severe venous hemorrhage and hepatic injury in swine. J Trauma. 2003;54:177-182.
2. Gustafson SB, Fulkerson P, et al. Chitosan dressing provides hemostasis in swine femoral arterial injury model. Prehospital emergency care. 2007;11: 172-178.
3. Wedmore I, McManus JG, et al. A special report on chitosan based hemostatic dressing: Experience in current combat operations. J Trauma. 2006;60:655- 658 .

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years old
* Signing an informed consent
* Percutaneous coronary angiography with a 6 french sheath via the femoral artery
* Post catheterization non-invasive systolic blood pressure 150 mm Hg

Exclusion criteria:

* STEMI
* Patients who received IIb-IIIa antagonists before or during angiography.
* Patients who received more than 2500u IV Heparin or more than 0.5 mg/kg LMWH within 8 hours before the procedure.
* Known bleeding tendency, disturbed clotting system or platelet function
* Evidence of bleeding or hematoma at the access site prior to sheath removal.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Actual)
Dates: Start 2008-01; Primary Completion 2009-01 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Primary efficacy endpoint will be time to hemostasis. | 1 hour

SECONDARY OUTCOMES:
be safety (complication rate) and satisfaction of patients regarding time to sitting incline and time to ambulation. 25% of patients from each arm will be randomized for Duplex examination of the femoral artery at the access site. | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Morris Mosseri, MD, Principal Investigator — Tel-Aviv University, Sackler School of Medicine
Locations (1):
- Meir Medical Center, Kfar Saba, Israel

REFERENCES:
- [Background] Wedmore I, McManus JG, Pusateri AE, Holcomb JB. A special report on the chitosan-based hemostatic dressing: experience in current combat operations. J Trauma. 2006 Mar;60(3):655-8. doi: 10.1097/01.ta.0000199392.91772.44. PMID 16531872
- [Background] Pusateri AE, McCarthy SJ, Gregory KW, Harris RA, Cardenas L, McManus AT, Goodwin CW Jr. Effect of a chitosan-based hemostatic dressing on blood loss and survival in a model of severe venous hemorrhage and hepatic injury in swine. J Trauma. 2003 Jan;54(1):177-82. doi: 10.1097/00005373-200301000-00023. PMID 12544915
- [Background] Gustafson SB, Fulkerson P, Bildfell R, Aguilera L, Hazzard TM. Chitosan dressing provides hemostasis in swine femoral arterial injury model. Prehosp Emerg Care. 2007 Apr-Jun;11(2):172-8. doi: 10.1080/10903120701205893. PMID 17454803